CLINICAL TRIAL: NCT02679508
Title: Vonoprazan Study In Patients With Erosive Esophagitis to Evaluate Long-term Safety: A Study to Evaluate the Safety of Long-term Administration of Vonoprazan in Maintenance Treatment in Patients With Erosive Esophagitis (EE)
Brief Title: Vonoprazan Study in Patients With Erosive Esophagitis to Evaluate Long-term Safety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vonoprazan-4003; U1111-1178-8948 (Registry Identifier: WHO); JapicCTI-163153 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Erosive Esophagitis
Keywords: Esophagitis
MeSH Terms: conditions — Esophagitis | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan group (Experimental): Vonoprazan 20 mg administered orally once daily in the healing phase + vonoprazan 10 mg (as the initial dose and adjusted to vonoprazan 10 mg or 20 mg) administered orally once daily in the maintenance phase
  Interventions: Drug: Vonoprazan
- Lansoprazole group (Active Comparator): Lansoprazole 30 mg administered orally once daily in the healing phase + lansoprazole 15 mg (as the initial dose and adjusted to lansoprazole 15 mg or 30 mg) administered orally once daily in the maintenance phase
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan fumarate 10 mg or 20 mg capsules
  Arms: Vonoprazan group
Drug: Lansoprazole — Lansoprazole 15 mg or 30 mg capsules
  Arms: Lansoprazole group

SUMMARY:
The purpose of this study is exploratorily evaluate the effect on gastric mucosal tissue and the safety of long-term administration (260 weeks: 5 years) of vonoprazan 10 mg or 20 mg in patients receiving maintenance treatment after healed erosive esophagitis (EE), and the curative effect of vonoprazan 20 mg versus lansoprazole in patients with EE.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, parallel-group study to exploratorily evaluate the effect on gastric mucosal tissue and the safety of long-term administration of vonoprazan in maintenance treatment after healed EE, and the curative effect of vonoprazan versus lansoprazole in participants with EE.

Participants endoscopically diagnosed with EE of Los Angeles (LA) Classification Grades A to D at the start of treatment (Week 0 of the healing phase) will be randomly assigned to receive either vonoprazan 20 mg or lansoprazole 30 mg to be taken once daily for up to 8 weeks. Subjects with healed EE as confirmed endoscopically at Week 4 or 8 in the healing phase will enter the maintenance phase.

In the maintenance phase, the vonoprazan group and the lansoprazole group will be administered a starting dose of 10 mg and 15 mg, respectively, once daily up to 260 weeks.

If the principal investigator or investigator judged the effect of vonoprazan 10 mg or lansoprazole 15 mg to be insufficient as the maintenance treatment of EE, vonoprazan and lansoprazole may be increased to 20 mg and 30 mg, respectively.

The research period will consist of two subperiods: healing phase in which participants with EE will receive treatment (for 4 or 8 weeks) and maintenance phase in which participants will receive maintenance treatment (for 260 weeks), and thus, a total of up to 268 weeks. The number of visits will be a maximum of 18 visits. Planned number of research subjects, as the number of research subjects for entry to the maintenance phase, will be 130 participants in the vonoprazan group and 65 participants in the lansoprazole group.

ELIGIBILITY:
Inclusion Criteria

Healing Phase:

1. Participants endoscopically diagnosed with EE of grades A to D by the LA Classification Grading System at the start of treatment (Week 0 of the healing phase)
2. Participants with H. pylori negative
3. Participants who, in the opinion of the principal investigator or investigator, are capable of understanding the content of the clinical research and complying with the research protocol requirements.
4. Participants who can sign and date an informed consent form and information sheet prior to the conduction of the clinical research procedures.
5. Male or female participants aged 20 years or older at the time of informed consent
6. Therapeutic category: Ambulatory

   Maintenance Phase:
7. Participants who have endoscopically confirmed EE healing* (mucous membrane disorder is not observed) at completion of the healing phase (Week 4 or 8 of the healing phase)

   * Participants who are classified as grade 0 according to severity classification of EE (See Table 9.b)
8. Participants who have been determined to be appropriate as subjects for maintenance treatment of EE by the principal investigator or investigator

Exclusion Criteria:

Healing Phase:

1. Participants with concurrent peptic ulcer (except scarred stage) or Zollinger-Ellison syndrome
2. Participants who received treatment with PPIs (including vonoprazan) within 4 weeks (Week -4 to Week 0) prior to the start of healing phase (Week 0 of the healing phase)
3. Participants with a history of H. pylori eradication.
4. Participants who have received surgery or treatment affecting gastroesophageal reflux (fundoplication or dilation for esophageal stenosis [excluding Schatzki's ring], etc.)
5. Participants with an esophagus-related complication (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal stenosis, etc.), a history of radiotherapy or cryotherapy of the esophagus, a caustic or physiochemical trauma (esophageal sclerotherapy, etc.). However, participants with Schatzki's ring (mucosal tissue ring around inferior esophageal sphincter) or Barrett's esophagus are allowed to be included.
6. Participants with clinically apparent hepatic impairment (e.g., AST or ALT levels at the time of informed consent: >1.5 times the upper limit of normal (ULN).
7. Participants with renal impairment or renal failure [creatinine clearance (CCr) ˂30 mL/min, etc.]
8. Participants with a history of hypersensitivity or allergy for PPIs.
9. Participants with a history of gastrectomy, gastrointestinal resection, or vagotomy
10. Participants with a malignant tumor
11. Participants who are pregnant, breast-feeding, possibly pregnant, or planning to become pregnant
12. Participants with one of the diseases listed under administration contraindication in the vonoprazan or lansoprazole package insert
13. Participants planning to take prohibited concomitant medications during the research period
14. Participants participating in other clinical studies
15. Participants who have been determined to be inappropriate as subjects in the study by the principal investigator or investigator

    Maintenance Phase:
16. Participants who have taken PPIs other than the study drug or the control drug during the healing phase
17. Participants who have been determined to be inappropriate as subjects in the study by the principal investigator or investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-03-20 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (36):
- Japan (36):
  - Tokatsu Tsujinaka Hospital, Abiko, Chiba
  - Hohnodai Hospital National Center For Global Health and Medicine, Ichikawa, Chiba
  - Red Cross Matsuyama Hospital, Matsuyama, Ehime
  - Kawakubo Clinic, Kama, Fukuoka
  - Hakodate Hospital, Hakodate, Hokkaido
  - Aoyama Medical Clinic, Kobe, Hyōgo
  - Hyogo College Of Medicine, Nishinomiya, Hyōgo
  - KKR Takamatsu Hospital, Takamatsu, Kagawa-ken
  - Shirane Clinic, Sendai, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - Shin-Beppu Hospital, Beppu, Oita Prefecture
  - Kawasaki Medical University, Kurashiki, Okayama-ken
  - Shiga Hospital, Ōtsu, Shiga
  - Shiga University Of Medical Science Hospital, Ōtsu, Shiga
  - Shimane University Hospital, Izumo, Shimane
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - Kohga Hospital, Yaizu, Shizuoka
  - Masuyama Clinic, Ōtawara, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Banno Clinic, Ōta-ku, Tokyo
  - Shimokitazawa Tomo Clinic, Setagaya-ku, Tokyo
  - National Center For Global Health and Medicine, Shinjyuku-ku, Tokyo
  - Nippon Medical School Hospital, Shinjyuku-ku, Tokyo
  - Chihaya Hospital, Fukuoka
  - Harada Hospital, Fukuoka
  - Kimura Shiro Clinic, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Mori Clinic, Fukuoka
  - Hanabata Clinic, Kumamoto
  - Morinaga Ueno Clinic, Kumamoto
  - Oki Hospital, Kyoto
  - Asahigaoka Hospital, Okayama
  - Kawasaki Hospital, Okayama
  - Arita Hospital, Ōita
  - Matsuki Clinic, Shizuoka
  - Oizumi Medical Clinic, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Uemura N, Kinoshita Y, Haruma K, Kushima R, Yao T, Akiyama J, Aoyama N, Baba Y, Suzuki C, Ishiguro K. Vonoprazan as a Long-term Maintenance Treatment for Erosive Esophagitis: VISION, a 5-Year, Randomized, Open-label Study. Clin Gastroenterol Hepatol. 2025 Apr;23(5):748-757.e5. doi: 10.1016/j.cgh.2024.08.004. Epub 2024 Aug 27. PMID 39209187
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603a4db2bf003ab4a26b

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 36 investigative sites in Japan, from 20 March 2016 to 5 March 2022.
Pre-assignment Details: Participants with a historical diagnosis of erosive esophagitis were enrolled. Participants received Vonoprazan or Lansoprazole as part of a routine medical care.
Groups:
- Vonoprazan Group: Vonoprazan 20 mg administered orally once daily in the healing phase, after that Vonoprazan 10 mg (as the initial dose and adjusted to Vonoprazan 10 mg or 20 mg) administered orally once daily in the maintenance phase.
- Lansoprazole Group: Lansoprazole 30 mg administered orally once daily in the healing phase, after that Lansoprazole 15 mg (as the initial dose and adjusted to Lansoprazole 15 mg or 30 mg) administered orally once daily in the maintenance phase.
Period: Healing Phase
Arm/Group | Vonoprazan Group | Lansoprazole Group
Started | 139 | 69
Completed | 137 | 68
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Maintenance Phase
Arm/Group | Vonoprazan Group | Lansoprazole Group
Started | 137 | 68
Completed | 105 | 53
Not Completed | 32 | 15
Not completed — Adverse Event | 12 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 15 | 8
Not completed — Other | 5 | 4

BASELINE CHARACTERISTICS:
Population: Randomized Set: All participants who were enrolled in Healing Phase and who received at least one dose of any therapy during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vonoprazan Group | Lansoprazole Group | Total
Number analyzed (Participants) | 139 | 69 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (11.90) | 61.8 (12.13) | 60.9 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 27 | 68
  Male | 98 | 42 | 140
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 139 | 69 | 208
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 164.4 (8.96) | 162.7 (10.12) | 163.8 (9.37)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 68.55 (13.011) | 65.98 (11.520) | 67.70 (12.566)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2]
  Kilogram (kg)/meter (m)^2 | 25.25 (3.737) | 24.85 (3.280) | 25.12 (3.589)
Smoking History [Count of Participants; unit: Participants]
  Never Smoked | 52 | 31 | 83
  Current Smoker | 25 | 9 | 34
  Ex-Smoker | 62 | 29 | 91
Drinking History [Count of Participants; unit: Participants]
  Drinks Every Day | 44 | 17 | 61
  Drinks a Few Days per Week | 27 | 16 | 43
  Drinks a Few Days per Month | 22 | 19 | 41
  Never Drank or Ex Drinker | 46 | 17 | 63
Consumption of Caffeine-Containing Beverage [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Consume caffeine-containing beverage almost everyday?" were reported.
  Participants
    Yes | 112 | 50 | 162
    No | 27 | 19 | 46
Endoscopic Findings in Esophagus [Count of Participants; unit: Participants] — Endoscopic findings were assessed using the Los Angeles (LA) classification. The LA classification graded as follows- Grade O: normal mucosa; Grade A: nonconfluent mucosal breaks <5 mm in length; Grade B: nonconfluent mucosal breaks ≥ 5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential.
  Participants
    Grade A | 64 | 33 | 97
    Grade B | 50 | 25 | 75
    Grade C | 20 | 10 | 30
    Grade D | 5 | 1 | 6
Serum Gastrin Level [Mean (Standard Deviation); unit: Picogram/milliliter (pg/mL)] | 130.2 (77.97) | 155.1 (128.73) | 138.5 (98.15)
Serum Pepsinogen I/II Ratio [Mean (Standard Deviation); unit: Ratio] — Serum Pepsinogen I/II ratio for each group were reported. The Serum Pepsinogen I/II ratio was calculated by concentration of Pepsinogen I in serum divided by concentration of Pepsinogen II in serum *100.
  Ratio | 5.45 (1.226) | 5.24 (1.314) | 5.38 (1.257)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Malignant Alteration of Epithelial Cells
Description: Numbers of participants with malignant alteration of epithelial cells for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for gastric mucosa histopathology. The number analyzed is the number of participants with data available for analysis.
Time Frame: Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: Safety Data Analysis Set in the Maintenance Phase: All participants who were enrolled in Maintenance Phase and who received at least one dose of any therapy in the Maintenance Phase of this study. The number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Parietal Cell Protrusion/Hyperplasia
Description: Numbers of participants with parietal cell protrusion/hyperplasia for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for gastric mucosa histopathology. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 99 | 45

3. Primary Outcome: Number of Participants With Foveolar Hyperplasia
Description: Numbers of participants with foveolar hyperplasia for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for gastric mucosa histopathology. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 15 | 1

4. Primary Outcome: Number of Participants With Enterochromaffin-like-cell Hyperplasia
Description: Numbers of participants with enterochromaffin-like-cell hyperplasia for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for gastric mucosa histopathology. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 5 | 4

5. Primary Outcome: Number of Participants With G-cell Hyperplasia
Description: Numbers of participants with G-cell hyperplasia for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for gastric mucosa histopathology. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 87 | 40

6. Secondary Outcome: Percentage of Participants With Recurrence of Erosive Esophagitis (EE)
Description: Erosive esophagitis recurrence is defined as endoscopically confirmed to have erosive esophagitis (LA classification grades O and A to D) during the Maintenance Phase. The LA classification graded as follows- Grade O: normal mucosa; Grade A: nonconfluent mucosal breaks <5 mm in length; Grade B: nonconfluent mucosal breaks ≥ 5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: Full Analysis Set in the Maintenance Phase: All participants who were randomized and who received at least one dose of any therapy in the Maintenance Phase of this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 135 | 67
Percentage of participants | 3.8 [1.1 to 9.6] | 11.3 [4.3 to 23.0]

7. Secondary Outcome: Percentage of Participants Who Healed EE at the End of Healing Phase
Description: Percentage of participants who healed EE at the end of healing phase was reported.
Time Frame: Up to Week 8
Population: Full Analysis Set in the Healing Phase: All participants who were randomized and who received at least one dose of any therapy in the Healing Phase of this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 139 | 69
Percentage of participants | 1.4 [0.2 to 5.1] | 0.0 [0.0 to 5.2]

8. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) in Maintenance Phase
Description: Number of participants reporting one or more TEAEs in Maintenance Phase was reported. An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: 260 weeks (Baseline, up to the end of Maintenance Phase)
Population: Safety Data Analysis Set in the Maintenance Phase: All participants who were enrolled in Maintenance Phase and who received at least one dose of any therapy in the Maintenance Phase of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 135 | 67
Participants | 126 | 64

9. Secondary Outcome: Number of Participants With Fundic Gland Polyp
Description: Numbers of participants with fundic gland polyp for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for endoscopic findings. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 104 | 53
Participants | 75 | 45

10. Secondary Outcome: Number of Participants With Hyperplastic Polyp
Description: Numbers of participants with hyperplastic polyp for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for endoscopic findings. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 104 | 53
Participants | 24 | 6

11. Secondary Outcome: Number of Participants With Cobblestone Mucosa
Description: Numbers of participants with cobblestone mucosa for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for endoscopic findings. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 104 | 53
Participants | 23 | 8

12. Secondary Outcome: Number of Participants With Multiple White and Flat Elevated Lesions
Description: Numbers of participants with multiple white and flat elevated lesions for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for endoscopic findings. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 104 | 53
Participants | 8 | 9

13. Secondary Outcome: Number of Participants With Black Spots
Description: Numbers of participants with black spots for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as the endpoint for endoscopic findings. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 104 | 53
Participants | 8 | 7

14. Secondary Outcome: Number of Participants With Inflammation (Mononuclear Infiltration) in Greater Curvature of Middle Gastric Body
Description: Numbers of participants with inflammation (mononuclear infiltration) in greater curvature of the middle gastric body for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 15 | 9

15. Secondary Outcome: Number of Participants With Inflammation (Mononuclear Infiltration) in Greater Curvature of Antrum
Description: Numbers of participants with inflammation (mononuclear infiltration) in greater curvature of the antrum for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 11 | 9

16. Secondary Outcome: Number of Participants With Neutrophilic Infiltration in Greater Curvature of Middle Gastric Body
Description: Numbers of participants with neutrophilic infiltration in greater curvature of the middle gastric body for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 1 | 0

17. Secondary Outcome: Number of Participants With Neutrophilic Infiltration in Greater Curvature of Antrum
Description: Numbers of participants with neutrophilic infiltration in greater curvature of the antrum for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 0 | 0

18. Secondary Outcome: Number of Participants With Atrophy in Greater Curvature of Middle Gastric Body
Description: Numbers of participants with atrophy in greater curvature of the middle gastric body for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 0 | 0

19. Secondary Outcome: Number of Participants With Atrophy in Greater Curvature of Antrum
Description: Numbers of participants with atrophy in greater curvature of the antrum for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 7 | 7

20. Secondary Outcome: Number of Participants With Intestinal Metaplasia in Greater Curvature of Middle Gastric Body
Description: Numbers of participants with intestinal metaplasia in greater curvature of the middle gastric body for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With Intestinal Metaplasia in Greater Curvature of Antrum
Description: Numbers of participants with intestinal metaplasia in greater curvature of the antrum for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 6 | 6

22. Secondary Outcome: Number of Participants With Presence of H.Pylori in Greater Curvature of Middle Gastric Body
Description: Numbers of participants with presence of H.pylori in greater curvature of the middle gastric body for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 0 | 0

23. Secondary Outcome: Number of Participants With Presence of H.Pylori in Greater Curvature of Antrum
Description: Numbers of participants with presence of H.pylori in greater curvature of the antrum for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported as histological assessment of gastritis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 102 | 52
Participants | 0 | 0

24. Secondary Outcome: Number of Participants With Gastric Polyp
Description: Numbers of participants with gastric polyp for Vonoprazan group and Lansoprazole group at Week 268 (Week 260 in Maintenance Phase) were reported. The number analyzed is the number of participants with data available for analysis.
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan Group | Lansoprazole Group
Number analyzed (Participants) | 104 | 53
Participants | 82 | 46

ADVERSE EVENTS:
Time Frame: Up to Week 268 (Week 260 in Maintenance Phase)
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Vonoprazan Group | Lansoprazole Group
All-Cause Mortality (participants affected / at risk) | 0/139 | 1/69
Serious Adverse Events (participants affected / at risk) | 50/139 | 27/69
Other Adverse Events (participants affected / at risk) | 128/139 | 65/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan Group (N=139) | Lansoprazole Group (N=69)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 3 | 6
Cataract nuclear (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 5 | 4
Inguinal hernia (Gastrointestinal disorders) | 2 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 3 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatic steatosis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholangitis infective (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to retroperitoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 3 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 1 | 0
Peripheral nerve palsy (Nervous system disorders) | 1 | 0
Sciatic nerve palsy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan Group (N=139) | Lansoprazole Group (N=69)
Vertigo (Ear and labyrinth disorders) | 7 | 1
Gastric polyps (Gastrointestinal disorders) | 62 | 31
Gastric mucosal lesion (Gastrointestinal disorders) | 30 | 17
Gastritis erosive (Gastrointestinal disorders) | 12 | 9
Diarrhoea (Gastrointestinal disorders) | 13 | 6
Large intestine polyp (Gastrointestinal disorders) | 11 | 6
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 10 | 6
Constipation (Gastrointestinal disorders) | 8 | 4
Dental caries (Gastrointestinal disorders) | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 4
Nasopharyngitis (Infections and infestations) | 49 | 29
Bronchitis (Infections and infestations) | 13 | 7
Influenza (Infections and infestations) | 13 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 6
Gastroenteritis (Infections and infestations) | 8 | 4
Cystitis (Infections and infestations) | 8 | 2
Pharyngitis (Infections and infestations) | 5 | 5
Herpes zoster (Infections and infestations) | 3 | 4
Tonsillitis bacterial (Infections and infestations) | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 8 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Headache (Nervous system disorders) | 6 | 4
Dizziness (Nervous system disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 7 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Eczema (Skin and subcutaneous tissue disorders) | 10 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 4
Hypertension (Vascular disorders) | 15 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT02679508/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT02679508/SAP_001.pdf